CLINICAL TRIAL: NCT04541394
Title: Effectiveness and Clinical Application of MolecuLight Bacterial Fluorescence Imaging in Wound Debridement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chang shun cheng, Director of Wound Care Center and Department of Plastic Surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202006059
Record Dates: First submitted 2020-08-11; First posted 2020-09-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Infection, Surgical Site
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MolecuLight group (Experimental): Patients with infected wounds received MolecuLight photography during debridement operation to evaluate the adequacy of remission of infected biofilm and facilitate wound healing
  Interventions: Device: MolecuLight
- Control group (No Intervention): Patients with infected wounds received debridement operation by surgeon's clinical experiences to decide the extension of wounds

INTERVENTIONS:
Device: MolecuLight — MolecuLight is a device that utilizes a special light which, when used on wounds, helps identify the regions which pathogenic bacterial counts are the highest. The device applies 405nm violet light which is harmless to the human tissue. When specific components in bacteria catches up the light, a photoluminescent reaction is triggered and the fluorescence light is caught by the camera on this device in real time.
  Arms: MolecuLight group

SUMMARY:
MolecuLight is a device that utilizes a special light which, when used on wounds, helps identify the regions which pathogenic bacterial counts are the highest. The device applies 405nm violet light which is harmless to the human tissue. When specific components in bacteria catches up the light, a photoluminescent reaction is triggered and the fluorescence light is caught by the camera on this device in real time.

When treating an infected wound which requires debridement and/or reconstruction, traditionally surgeons rely on many clinical clues to judge the severity and region of infection. However, these clues, such as lab data, vital signs, bacterial culture growth, or infection symptoms/signs, are usually indirect and also require several days to be fully interpretated.

The advantage of MolecuLight is its simple, direct, real-time, and flexible application, which is very important and valuable when treating an infected wound. We aim to add this device to our routines and see if the treatment course for these wounds can be more rapid and effective, and also utilize the countless potential of immediate bacterial identification in numerous aspects of our work.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wounds that present obvious symptoms or/and signs of infection, and chronic wounds that have failed to heal or improve for 14 days (Chronic wounds are often complicated or caused by wound infection)
* Patients that are scheduled for surgical treatment for the wound
* Patients that are older than (including) 20 years and younger than (including) 85 years.
* Wounds with a size larger than 1x1 cm2

Exclusion Criteria:

* Wounds that heal within 14 days.
* Patient is unable to continue further surgical treatment due to any reason
* The wound site is amputated
* Patient refuses further surgical treatment
* The patient has an active malignancy currently under treatment
* Patient is immunocompromised or currently under systemic steroid treatment
* The wound had been treated by radiation
* The patient refuses to participate in this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of residual bacterial light spots | Immediately after each debridement within surgery
  The percentage of residual bacterial light spots. After each debridement, we use MolecuLight to evaluate the residual shinny area (post-debridement shinny area/pre-debridement shinny area)
Numbers of Re-debridement | Immediately after each surgery
  If the bacterial shinny area after debridement > 10% wound area, the debridement will be performed again until < 10% residual bacterial shinny area
Duration of wound healing | Time of complete epithelialization without drainage
  Time of complete epithelialization without drainage

SECONDARY OUTCOMES:
Incidence of surgical complications | 8 weeks postoperatively
  Incidence of wound bleeding, infection and necrosis after debridement
Antibiotic use | 8 weeks postoperatively
  The amount (regimen and dosage)
Duration of antibiotic use | 8 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Shun Cheng Chang, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital First Medical Building, New Taipei City, Taiwan